CLINICAL TRIAL: NCT05449249
Title: Oral and Gut Microbiota Changes During Long-term Fasting in Humans
Acronym: OralFast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buchinger Wilhelmi Development & Holding GmbH (Other)
Collaborators: Buchinger Wilhelmi Clinic (Unknown); University of Geneva, Switzerland (Other); King's College London (Other); ETH Zurich (Switzerland) (Other)
Responsible Party: Principal Investigator, Françoise Wilhelmi de Toledo, Scientific Director; Principal Investigator, Buchinger Wilhelmi Development & Holding GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BuWi_OralFast_2022
Record Dates: First submitted 2022-06-29; First posted 2022-07-08 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Healthy; Periodontitis
Keywords: oral microbiota; intestinal microbiota; inflammatory status; redox status; sulfur metabolism; halitosis
MeSH Terms: conditions — Periodontitis; Halitosis

STUDY DESIGN:
Intervention Model Description: single-arm, prospective, monocentric, interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Long-term fasting (Experimental): Long-term fasting according to the Buchinger Wilhelmi fasting program.
  Interventions: Procedure: Long-term fasting

INTERVENTIONS:
Procedure: Long-term fasting — The participants will undergo a fasting program that includes the daily intake of 250 kcal under medical supervision.

SUMMARY:
The aim of this longitudinal trial is to investigate the effects of a 10±3-day fasting period in 30 subjects. Changes in the oral and gut microbiota, halitosis, as well as inflammatory and antioxidative parameters and biomarkers of sulfur metabolism will be analysed.

DETAILED DESCRIPTION:
Fasting has been linked with changes in gut microbiota as part of the physiological adaptation. Furthermore, associations have been described between oral disease and nutrition (diet rich in carbohydrates). The aim of the present longitudinal clinical study is to explore the effect of a 10±3-day fasting period on the oral and gut microbiota. 30 systemically healthy subjects attending the Buchinger Wilhelmi Clinics for fasting, will participate. Changes in oral microbiota will be assessed in plaque and saliva samples and a number of inflammatory markers will be analyzed in Gingival Crevicular fluid (GCF) and blood obtained before, during and after the fasting period. The changes in the oral microbiota will be associated to the composition of the gut microbiota. Changes in periodontal parameters and halitosis related to the fasting period will be further evaluated. Given the known association between sulfur metabolism and the redox status, parameters from the antioxidant status and oxidative damages will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Both subjects with periodontitis and healthy periodontium will be included.
* Signed informed consent

Exclusion Criteria:

* Not able to sign the informed consent
* diagnosticated with cachexia, anorexia, nervosa, advanced kidney, liver or cerebrovascular insufficiency
* Smoking
* the intake of antibiotics within the last 8 weeks, as well as the intake of probiotics within the last 4 weeks
* periodontal treatment in the last 6 months
* chronic manifest psychical and psychiatric diseases
* participation in another study
* pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-08 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Changes in halitosis | daily from baseline to the 3rd day of food reintroduction
  Concentration of volatile sulfide compounds (hydrogen sulfide, methylmercaptan and dimethyl sulphide) using the OralChrome devise
Changes in microbiota compositions of subgingival microbial and plaque sampling | Baseline, fasting day 10, food reintroduction day 3
  Aggregatibacter actinomycetemcomitans (Aa), Porphyromonas (Pg), Tannerella forsythia (Tf), Treponema denticola (Td), Parvimonas micra (Pm) and Prevotella intermedia (Pi) analysed by RT-q-PCR
Changes in microbiota composition in saliva | Baseline, fasting day 10, food reintroduction day 3, 1 and 3 months afterwards
  16 rRNA gene amplicon sequencing
Changes in microbiota composition in faeces | Baseline, first spontaneous stool after food reintroduction (up to day 3), 1 and 3 months afterwards
  16 rRNA gene amplicon sequencing
Changes in total antioxidant capacity (TAC) | Baseline, fasting day 3, 5, 10
  (mmol DPPH/L)
Changes in hydrogen sulfide production capacity | at the beginning and the end of fasting, on day 3 and 5, as well as at the food reintroduction
  measured in serum and urine using the lead acetate assay

SECONDARY OUTCOMES:
Changes in glutathione (GSH) | Baseline, fasting day 3, 5, 10
  (µmol/g Hb)
Changes in thiobarbituric acid reactive substances (TBARS) | Baseline, fasting day 3, 5, 10
  (µmol/L)
Changes in malondialdehyde (MDA) | Baseline, fasting day 3, 5, 10
  nM/L
Changes in protein carbonyls | Baseline, fasting day 3, 5, 10
  (nmol/mg protein)
Changes in nicotinamide adenine dinucleotide phosphate (NADPH) oxidase | Baseline, fasting day 3, 5, 10
  (µL)
Changes in glutathione reductase (GR) activity | Baseline, fasting day 3, 5, 10
  (U/g Hb)
Changes in glutathione peroxidase (GPx) activity | Baseline, fasting day 3, 5, 10
  (U/g Hb)
Changes in peroxiredoxin activity | Baseline, fasting day 3, 5, 10
  (U/g Hb)
Changes in catalase (CAT) activity | Baseline, fasting day 3, 5, 10
  (U/mg Hb)
Changes in superoxide dismutase (SOD) activity | Baseline, fasting day 3, 5, 10
  (U/g Hb)
Changes in hydroxyl radical scavenging | Baseline, fasting day 3, 5, 10
  (mmol deoxyribose/ml)
Changes in superoxydradical scavenging | Baseline, fasting day 3, 5, 10
  (mmol NBT/L plasma)
Changes in ABTS scavenging | Baseline, fasting day 3, 5, 10
  (mmol/L)
Changes in reducing power | Baseline, fasting day 3, 5, 10
  (mmol/L plasma)
Changes in thiosulfate | Baseline, fasting day 10, food reintroduction day 3
  measured using the monobromobimane method using HPLC and LC-MS/MS
Changes in persulfidation | Baseline, fasting day 10, food reintroduction day 3
  persulfidation in serum and urine
Changes in cystein | Baseline, fasting day 10, food reintroduction day 3
  using the S-sulfocysteine (SSC) method which is a HPLC-based method using automated precolumn derivatization with OPA and UV detection at 338 nm in serum and urine
Changes in amino acid metabolites | Baseline, fasting day 10, food reintroduction day 3
  using a targeted approach in serum and urine
Changes in IL-10 in blood | Baseline, fasting day 10, food reintroduction day 3
  analysed in blood with Bio-Plex 200 Suspension array System
Changes in G-CSF in blood | Baseline, fasting day 10, food reintroduction day 3
  analysed in blood with Bio-Plex 200 Suspension array System
Changes in IFN-γ in blood | Baseline, fasting day 10, food reintroduction day 3
  analysed in blood with Bio-Plex 200 Suspension array System
Changes in TNF-α in blood | Baseline, fasting day 10, food reintroduction day 3
  analysed in blood with Bio-Plex 200 Suspension array System
Changes in IL-1β in blood | Baseline, fasting day 10, food reintroduction day 3
  analysed in blood with Bio-Plex 200 Suspension array System
Changes in IL-6 in blood | Baseline, fasting day 10, food reintroduction day 3
  analysed in blood with Bio-Plex 200 Suspension array System
Changes in IL-8 in blood | Baseline, fasting day 10, food reintroduction day 3
  analysed in blood with Bio-Plex 200 Suspension array System
Changes in IL-17 in blood | Baseline, fasting day 10, food reintroduction day 3
  analysed in blood with Bio-Plex 200 Suspension array System
Changes in IL-10 in gingival crevicular fluid | Baseline, fasting day 10, food reintroduction day 3
  analysed in gingival crevicular fluid with Bio-Plex 200 Suspension array System
Changes in G-CSF in gingival crevicular fluid | Baseline, fasting day 10, food reintroduction day 3
  analysed in gingival crevicular fluid with Bio-Plex 200 Suspension array System
Changes in IFN-γ in gingival crevicular fluid | Baseline, fasting day 10, food reintroduction day 3
  analysed in gingival crevicular fluid with Bio-Plex 200 Suspension array System
Changes in TNF-α in gingival crevicular fluid | Baseline, fasting day 10, food reintroduction day 3
  analysed in gingival crevicular fluid with Bio-Plex 200 Suspension array System
Changes in IL-1β in gingival crevicular fluid | Baseline, fasting day 10, food reintroduction day 3
  analysed in gingival crevicular fluid with Bio-Plex 200 Suspension array System
Changes in IL-6 in gingival crevicular fluid | Baseline, fasting day 10, food reintroduction day 3
  analysed in gingival crevicular fluid with Bio-Plex 200 Suspension array System
Changes in IL-8 in gingival crevicular fluid | Baseline, fasting day 10, food reintroduction day 3
  analysed in gingival crevicular fluid with Bio-Plex 200 Suspension array System
Changes in IL-17 in gingival crevicular fluid | Baseline, fasting day 10, food reintroduction day 3
  analysed in gingival crevicular fluid with Bio-Plex 200 Suspension array System

OTHER OUTCOMES:
Changes in Rosenberg scale | daily from baseline to the 3rd day of food reintroduction
  organoleptic intensity scale for measuring oral malodor: 0 = no odor to 5 = intense odor
Changes in Seemann scale | daily from baseline to the 3rd day of food reintroduction
  organoleptic assessment: 1 = odor noticable from 10 cm to 3 = odor noticeable from 1m
Changes in Ayurvedic diagnosis of the tongue | daily from baseline to the 3rd day of food reintroduction
  examination of the tongue
Changes in urinary ketone bodies | daily from baseline to the 3rd day of food reintroduction
  using ketostix
Changes in capillary blood ketones | daily from baseline to the 3rd day of food reintroduction
  using GlucoMen areo 2k
Changes in capillary blood glucose | daily from baseline to the 3rd day of food reintroduction
  using GlucoMen areo 2k
Changes in ph value of the urin | daily from baseline to the 3rd day of food reintroduction
  using test strips
Changes in weight | daily from baseline to the 3rd day of food reintroduction as well as 1 and 3 months after
  kg
Changes in blood pressure | daily from baseline to the 3rd day of food reintroduction as well as 1 and 3 months after
  systolic and diastolic in mmHg
Changes in pulse | daily from baseline to the 3rd day of food reintroduction as well as 1 and 3 months after
  beats per minute
Plaque Index score | baseline
  Sillness & Loe, 1964: from 0 = no plaque to 3 = abundant plaque along the gingival margin, interdental spaces filled with plaque
Gingival index score | baseline
  Löe & Sillness, 1963: from 0 = normal gingiva to 3 = severe inflammation
Probing pocket depth | baseline
  Bleeding on probing, recorded as present within 30 sec (1) or absent (0)
clinical attachment level | baseline
  distance between the cemento-enamel junction and the tip of the graduated steel
recession | baseline
  distance between CEJ and marginal edge of the free gingiva
Changes in leucocytes | Baseline, fasting day 10, and food reintroduction day 3
  (thousands/µl)
Changes in erythrocytes | Baseline, fasting day 10, and food reintroduction day 3
  (millions/µl)
Changes in haemoglobin | Baseline, fasting day 10, and food reintroduction day 3
  (g/dl)
Changes in haematocrit | Baseline, fasting day 10, and food reintroduction day 3
  (in %)
Changes in MCV | Baseline, fasting day 10, and food reintroduction day 3
  (fl)
Changes in MCH | Baseline, fasting day 10, and food reintroduction day 3
  (pg)
Changes in MCHC | Baseline, fasting day 10, and food reintroduction day 3
  (g/dl)
Changes in thrombocytes | Baseline, fasting day 10, and food reintroduction day 3
  (thousands/µl)
Changes in international normalized ratio | Baseline, fasting day 10, and food reintroduction day 3
  ratio
Changes in Quick | Baseline, fasting day 10, and food reintroduction day 3
  (in %)
Changes in partial thromboplastin time | Baseline, fasting day 10, and food reintroduction day 3
  (sec)
Changes in aspartate aminotransferase (AST/GOT) | Baseline, fasting day 10, and food reintroduction day 3
  (U/l)
Changes in alanine aminotransferase (ALT/GPT) | Baseline, fasting day 10, and food reintroduction day 3
  (U/l)
Changes in gamma-glutamyl transferase (GGT) | Baseline, fasting day 10, and food reintroduction day 3
  (U/l)
Changes in alkaline phosphatase | Baseline, fasting day 10, and food reintroduction day 3
  (U/l)
Changes in uric acid | Baseline, fasting day 10, and food reintroduction day 3
  (mg/dl)
Changes in urea | Baseline, fasting day 10, and food reintroduction day 3
  (mg/dl)
Changes in glomerular Filtration Rate (GFR) | Baseline, fasting day 10, and food reintroduction day 3
  (ml/min/1.73m2KOF)
Changes in creatinine | Baseline, fasting day 10, and food reintroduction day 3
  (mg/dl)
Changes in thyroid-stimulating hormone (TSH) | Baseline, fasting day 10, and food reintroduction day 3
  (mE/l)
Changes in total cholesterol | Baseline, fasting day 10, and food reintroduction day 3
  (mg/dl)
Changes in triglyceride | Baseline, fasting day 10, and food reintroduction day 3
  (mg/dl)
Changes in high-density lipoprotein (HDL) | Baseline, fasting day 10, and food reintroduction day 3
  (mg/dl)
Changes in low-density lipoprotein (LDL) | Baseline, fasting day 10, and food reintroduction day 3
  (mg/dl)
Changes in LDL / HDL - ratio | Baseline, fasting day 10, and food reintroduction day 3
  ratio
Changes in glucose | Baseline, fasting day 10, and food reintroduction day 3
  (mg/dl)
Changes in HbA1c | Baseline, fasting day 10, and food reintroduction day 3
  (mmol/mol)
Changes in sodium | Baseline, fasting day 10, and food reintroduction day 3
  (mmol/l)
Changes in potassium | Baseline, fasting day 10, and food reintroduction day 3
  (mmol/l)
Changes in calcium | Baseline, fasting day 10, and food reintroduction day 3
  (mmol/l)
Changes in magnesium | Baseline, fasting day 10, and food reintroduction day 3
  (mmol/l)
Changes in erythrocyte sedimentation rate | Baseline, fasting day 10, and food reintroduction day 3
  (mm/h)
Changes in C - reactive protein | Baseline, fasting day 10, and food reintroduction day 3
  (mg/l)
Changes in pH value of saliva | Baseline, fasting day 10, food reintroduction day 3, 1 and 3 months afterwards
  (mol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Wilhelmi de Toledo, MD, Principal Investigator — Buchinger Wilhelmi
Locations (1):
- Buchinger Wilhelmi clinic, Überlingen, Germany

IPD SHARING:
Plan to Share IPD: No